CLINICAL TRIAL: NCT00162344
Title: AceP-D: Non-invasive Assessment of Atypical Chest Pain in Patients With Diabetes
Brief Title: A Study of Stress Heart Imaging in Patients With Diabetes at Risk for Coronary Disease.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Qi Zhu, MD Sr. Medical Director, Lantheus Medical Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARDIOLITE-404
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Technetium Tc 99m Sestamibi

INTERVENTIONS:
Drug: Technetium Tc99m Sestamibi

SUMMARY:
The study is designed to see if stress heart imaging can be used as a screening exam in patients with diabetes and risk factors of developing of coronary artery disease and experiencing future cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* History of diabetes for at least 5 years, with a least 2 risk factors (i.e. hypertension, elevated cholesterol levels, history of or current smoker, obese, family history of heart disease) & atypical chest pain.

Exclusion Criteria:

* Typical chest pain being treated with medication, unable to exercise, previous confirmed heart disease

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2003-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Examine the prevalence of ischemic heart disease in population of patients with diabetes mellitus and atypical chest pain.

SECONDARY OUTCOMES:
Determine the accuracy of myocardial perfusion imaging (MPI) and exercise tolerance testing (ETT) for the detection of coronary artery disease (CAD) in a subset of patients undergoing clinically indicated coronary angiography.
Determine the relative value of ETT, Duke Treadmill Score (DTS), MPI, ejection fraction (EF), clinical risk factors, and C-Reactive Protein (CRP) values for identifying patients at risk for cardiac events.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rosenberg, MD, Principal Investigator — Bristol-Myers Squibb
Locations (12):
- United States (11):
  - Local Institution, Mission Viejo, California
  - Local Institution, Rancho Santa Fe, California
  - Local Institution, San Diego, California
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Detroit, Michigan
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Albany, New York
  - Local Institution, Roslyn, New York
  - Local Institution, Columbus, Ohio
  - Local Institution, Houston, Texas
- Local Institution, Montreal, Quebec, Canada